CLINICAL TRIAL: NCT00434265
Title: OBESITY, PHYSICAL INACTIVITY OR DIETARY FAT ? Role of Physical Activity in the Trafficking of Dietary Fatty Acids Varying in Length and Saturation Degree.
Brief Title: Obesity, Physical Inactivity or Dietary Fat ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: PRNA (INSERM/INRA) (Unknown); Fondation Coeur et Artères (Other); Centre National de la Recherche Scientifique, France (Other); Louis Pasteur University, Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3493
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Obesity; Exercise; Fat oxidation; Overweigh (IMC>25 and IMC<30)
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Physical Conditioning, Human

INTERVENTIONS:
Behavioral: Physical training

SUMMARY:
Obesity is the consequence of a chronic disequilibrium of fat balance. Genetic factors determine predisposition to obesity, but the most often mentioned idea is that environmental factors, such as a high-fat diet and a sedentary lifestyle, join to favour weight gain and explain the increased prevalence of obesity in our westernized societies. Since lipogenesis is negligible in humans, obesity represents the consequence of altered fat partitioning between oxidation and storage, likely due to a preferential directing of dietary fat towards adipose tissue and away from muscle. Interventions that favour partitioning of dietary fat towards muscle for oxidation might thus protect against weight gain. Exercise may be one kind of such intervention but the scant data on dietary fat metabolism does not allow clear conclusions, in particular in obese subjects. One question concerns the impact of the type of fat eaten: the effects of physical inactivity may vary according to the length and saturation degree of the fatty acids. We hypothesize that 1) physical activity of moderate intensity, independently of its effect on energy balance, will favor a preferential trafficking towards adipose tissue, will modify the expression of genes implicated in fat oxidation and storage and partly correct the abnormalities observed in obese subjects, 2) effects of physical activity vary according to the saturation degree of fat. Twelve obese subjects, aged 18 to 55, will undergo tests before and after 2 months of training at current recommendations to ascertain dietary fat partitioning using stable isotopes and to determine changes in gene expression with muscle and adipose tissue microbiopsies.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 55
* IMC >25 and <30 kg/m2 and waist circumference >102 cm
* Familial antecedents of obesity
* Physical inactivity (PAL<1.5, according to MOSPA-questionnaire and accelerometry)
* Acceptation of physical training and body weight control during the study

Exclusion Criteria:

* Any drug interfering with energetic or lipid metabolism
* Any contradiction to moderate physical training
* Diabetes or arterial hypertension treatment
* Any other pathology (cardiovascular, psychiatric, renal or hepatic disease, viral hepatitis or VIH)
* Consumption of more than 40 g alcohol per day
* Recent voluntary or involuntary weight modification (3kg the next three months)
* A recent trip outside France before and during stable isotope measures.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Proportion of fat oxidation induced by physical training, according to fat type (oleate vs palmitate)

SECONDARY OUTCOMES:
Variations of oleate and palmitate postprandial kinetic in different lipoprotein fractions
Expression of different muscle and adipose tissue genes

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Simon, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service des Explorations Fonctionelles Respiratoires et de l'Exercice - Hôpital Civil, Strasbourg
  - Service de Médecine Interne et de Nutrition - Hôpital de Hautepierre, Strasbourg

REFERENCES:
- [Result] Jacobi D, Perrin AE, Grosman N, Dore MF, Normand S, Oppert JM, Simon C. Physical activity-related energy expenditure with the RT3 and TriTrac accelerometers in overweight adults. Obesity (Silver Spring). 2007 Apr;15(4):950-6. doi: 10.1038/oby.2007.605. PMID 17426330